CLINICAL TRIAL: NCT06458413
Title: :Single-arm, Phase II Clinical Trial of Utidelone Capsule Plus Capecitabine (CAP) in Patients With Metastatic Breast Cancer
Brief Title: Utidelone Capsule Plus Capecitabine (CAP) for Metastatic Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Min Yan, MD (Other Government)
Collaborators: Beijing Biostar Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Min Yan, MD, Professor, Henan Cancer Hospital
Organization: Henan Cancer Hospital (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BG02-2402
Record Dates: First submitted 2024-06-10; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer Recurrent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-arm (Experimental): Patients with HER2-negative breast cancer were treated with Utidelone Capsule combined with Capecitabine tablets.
  Interventions: Drug: Utidelone Capsule Plus Capecitabine

INTERVENTIONS:
Drug: Utidelone Capsule Plus Capecitabine — Utidelone Capsule: 60mg/m2/d, once daily, oral on an empty stomach, continuously administered for 1-5 days; Capecitabine tablets: 1000mg/m2, twice a day (daily dose 2000mg/m2), once in the morning and once in the evening, taken orally within 30 minutes after meals, and continuously administered for 14 days from day 1 to day 14.
  Every 21 days is a cycle .

SUMMARY:
This study aims to investigate the efficacy and safety of utidelone capsule plus Capecitabine in the treatment of advanced breast cancer , and thus provides a new systemic treatment strategy for those patients.

This study was a single-arm, phase II study of patients with recurrent or metastatic HER2-negative breast cancer who had previously received chemotherapy regimens containing taxanes and/or anthracyclines were treated with a combination of utidelone capsules and capecitabine. The main objective was to explore the efficacy and safety of the combined regimen.

DETAILED DESCRIPTION:
Patients with recurrent or metastatic HER2 negative breast cancer who have previously received chemotherapy containing taxanes and/or anthracyclines will receive combined treatment with utidelone capsule and capecitabine. Utidelone Capsule: 60mg/m2/d, once daily, oral on an empty stomach, continuously administered for 1-5 days; Capecitabine tablets: 1000mg/m2, twice a day (daily dose 2000mg/m2), once in the morning and once in the evening, taken orally within 30 minutes after meals, and continuously administered for 14 days from day 1 to day 14. Every 21 days is a cycle until disease progression, intolerable adverse events occur, subjects voluntarily withdraw, or the researcher determines that medication must be terminated.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in this study, sign an informed consent form, have good compliance, and are willing to follow-up.
2. Female, aged ≥ 18 and ≤ 70 years, with an ECOG score of 0-1 and an expected survival time of ≥ 12 weeks.
3. The pathological and/or cytological diagnosis (based on the latest biopsy results) is HER2 negative recurrent or metastatic breast cancer, regardless of hormone receptor status (ER/PR positive or negative, but the hormone receptor status needs to be determined);
4. All patients have received at least paclitaxel and/or anthracycline as a treatment option;
5. All patients with prior treatment ≤ 3 lines (for those who progress during the neoadjuvant/adjuvant period or within 12 months after the end of the last treatment, it is considered as the first line, and no progress is counted as the number of lines); For HR+/HER2- breast cancer patients, they also need to have received the first line systemic CDK4/6 inhibitor+endocrine therapy before the disease progresses.
6. According to RECIST 1.1 standard, there is at least one measurable extracranial lesion present.
7. Within one week before enrollment, the blood routine examination was basically normal (no blood transfusion within two weeks, no use of drugs to increase white blood cells or platelets):

   Neutrophil count (ANC) ≥ 1.5 × 109/L; Platelet count (PLT) ≥ 90 × 109/L; Hemoglobin ≥ 9.0 g/dL.
8. Within one week before enrollment, the blood biochemistry test was basically normal (based on the normal values of each research center laboratory): Total bilirubin (TBIL) ≤ 1.5 x Upper limit of normal value (ULN) SGPT/ALT ≤ 3 × ULN (liver metastasis patients ≤ 5 × ULN); SGOT/AST ≤ 3 × ULN (liver metastasis patients ≤ 5 × ULN); The creatinine clearance rate (Ccr) is ≥ 50 ml/min (Cockcroft Gault formula).
9. No major organ dysfunction
10. Women with fertility must agree to use effective contraceptive methods during the study period and within 6 months after the last study medication. Women with fertility must have a negative blood or urine pregnancy test before enrollment.

Exclusion Criteria:

1. Other malignant tumors within the 5 years prior to enrollment, excluding cured cervical carcinoma in situ, basal cell carcinoma of the skin, papillary thyroid carcinoma without lymph node metastasis, or squamous cell carcinoma of the skin.
2. Those who meet the following conditions:

   1. Received systemic anti-tumor therapy within 2 weeks prior to enrollment, including but not limited to endocrine therapy, small molecule targeted therapy, anti-tumor traditional Chinese medicine, etc;
   2. Within the 4 weeks prior to enrollment, chemotherapy, targeted biological therapy or immunotherapy, other clinical investigational drugs, radiation therapy, or major organ surgery (excluding biopsy) or significant trauma have been received, or elective surgery is required during the trial period. Those who have undergone major surgeries;
   3. Received nitroso urea or mitomycin C within 6 weeks prior to enrollment;
3. Individuals who have previously received treatment with Utidelone injection.
4. Peripheral neuropathy CTCAE 5.0 grade evaluation ≥ 2.
5. Those who have received treatment with capecitabine or other drugs with an active ingredient of 5-fluorouracil (excluding those who relapse after more than 12 months of treatment).
6. Pregnant and lactating patients.
7. Adverse reactions from previous anti-tumor treatments have not yet recovered to CTCAE 5.0 grade ≤1 (excluding toxicity judged by researchers to have no safety risk for hair loss).
8. Accompanied by meningeal metastasis; Accompanied by uncontrollable brain metastases (researchers have determined that new asymptomatic brain metastases or those known to have stable brain metastases after treatment can be enrolled); Or uncontrollable bone metastasis, which refers to patients who have or have recently been at risk of fractures or have obvious symptoms or other critical situations.
9. Uncontrollable pleural effusion, pericardial effusion, or abdominal effusion.
10. Individuals with active infections who currently require systematic anti infection treatment.
11. Have a history of immunodeficiency, including HIV antibody testing positive, or have other acquired or congenital immunodeficiency diseases, or have a history of organ transplantation.
12. Individuals with active hepatitis B or hepatitis C; Known active syphilis infection.
13. Have a history of severe cardiovascular and cerebrovascular diseases, including but not limited to:

    Serious cardiac rhythm or conduction abnormalities, such as ventricular arrhythmias requiring clinical intervention, grade II-III atrioventricular block, etc; At rest, the average QTcF obtained from three 12 lead electrocardiogram examinations is>470ms; Acute coronary syndrome, congestive heart failure, aortic dissection, stroke, or other Grade 3 or higher cardiovascular events occurring within 6 months prior to the first administration; Hypertension that cannot be controlled clinically. Other researchers have identified high-risk heart diseases.
14. Uncontrolled diabetes patients.
15. Patients with active gastrointestinal ulcers.
16. Have a clear history of neurological or psychiatric disorders, including epilepsy or dementia.
17. Participate in another clinical trial or use other investigational treatments simultaneously.
18. Individuals known to be allergic to the investigational drug or any of its excipients.
19. The researchers believe that the subjects have a history of other serious systemic diseases or other reasons that make them unsuitable to participate in this trial.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-05 (Actual); Primary Completion 2025-06-05 (Estimated); Study Completion 2025-12-05 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate （ORR） | 18 months
  ORR is defined as the percentage of participants in the analysis population who have CR or PR per RECIST 1.1.

SECONDARY OUTCOMES:
Progression-Free Survival（PFS） | 18 months
  time from the first dose to disease progression or any-cause death
Disease Control Rate （DCR） | 18 months
  DCR is defined as the percentage of participants in the analysis population who have CR or PR or SD per RECIST 1.1.
Duration of response (DoR) | 18 months
  DOR is defined as the interval from response initiation (when either CR or PR is first determined) to progression or death, whichever occurs first.
Overall survival (OS) | 18 months
  time from the first dose of study drug to any-cause death
Treatment-related Adverse Event-TRAE | Until 28 days after the last dose of treatment
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Cancer hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after de-identification are available following article publication.
Supporting Information: Study Protocol
Time Frame: Three years from publication
Access Criteria: Please contact Central contact person by Email